CLINICAL TRIAL: NCT02873117
Title: Evaluation of the Potential Association Between 5α-reductase Inhibitors Prescription and Occurrence of High Grade Prostate Cancers
Acronym: CANARI
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC13_8911_CANARI
Record Dates: First submitted 2016-08-16; First posted 2016-08-19 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Benign Prostate Hyperplasia
Keywords: Benign prostate hyperplasia; 5 alpha reductase inhibitor; prostate cancer; Symptomatic; treated
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms | interventions — Prostatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 5 alpha reductase inhibitor
  Interventions: Other: Prostate biopsy, prostatectomy or prostate resection
- Any other drug for benign prostate hyperplasia
  Interventions: Other: Prostate biopsy, prostatectomy or prostate resection

INTERVENTIONS:
Other: Prostate biopsy, prostatectomy or prostate resection — Collection of prostate examination

SUMMARY:
This is a multicenter, cohort study based on medico-administrative data from pathology laboratory registries and drug reimbursement files (CNAM-TS).

DETAILED DESCRIPTION:
Identification process will be retrospective and prospective using medico-administrative data from all pathology laboratory registries in Brittany and drug reimbursement files for patients living in Brittany, France.

An extraction from drug reimbursement files of French health reimbursement agency (CNAM-TS) for patients living in Brittany, France will be performed on the following request: reimbursement of any pharmacologic treatment patented for symptomatic benign hyperplasia between January 1st 2010 and December 31st 2011, and no diagnosis of prostate cancer before December 31st, 2011. This extraction has to be done in 2013 to catch data as far as 2010 and will encompass health reimbursement for prostate examination. A second extraction will be done in 2014 to complete data from the end of 2013.

Secondly, identification of patients will use pathology laboratory registries, based on code for prostate examination (prostate biopsy, prostatectomy or prostate resection); involvement of all pathology laboratories in Brittany ensures completeness of collection of prostate examination results for the study period (January 1st, 2012 to December 31st, 2013). A list of patients will be recorded at each pathology laboratory level with date of birth, date of prostate examination, type of exam, results with Gleason score along with a study number on electronic file.

By January 2014, link to reimbursement file (that is data on all reimbursement within 3 years: 2009 to 2011 previously extracted from the French health reimbursement agency) will be done thanks to three key variables (date of birth, date of prostate examination, identification of pathology laboratory) and all data from all centers will set up into one global file.

This design will allow evaluation of association between 5-ARI and either high grade prostate cancer or low grade prostate as opposite association could be observed. In addition this design focuses on the target population, i.e. patients with symptomatic benign prostate hyperplasia, identified through reimbursement of drugs patented for symptomatic benign prostate hyperplasia.

ELIGIBILITY:
Inclusion Criteria:

* Men with a reimbursement of any pharmacologic treatment patented for symptomatic benign prostate hyperplasia between January 1st 2010 and December 31st 2011, affiliated to French health system and living in Brittany, France.

Exclusion Criteria:

* Prostate cancer with a date of diagnosis before December 31st, 2011, patients enrolled in surveillance program with scheduled prostate biopsy, patients not affiliated to French health system.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Men treated for benign prostate hyperplasia
Sampling Method: Probability Sample
Enrollment: 5154 (Actual)
Dates: Start 2014-12; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
High grade (Gleason >= 7) prostate cancer | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Rennes, Rennes, France